CLINICAL TRIAL: NCT03224481
Title: Evaluation of the Effect of Tailored Electronic Reminders on Compliance With Removable Orthodontic Retention: A Randomised Controlled Trial
Brief Title: Evaluation of Tailored Electronic Reminders on Compliance With Removable Orthodontic Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11153
Record Dates: First submitted 2016-10-24; First posted 2017-07-21 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Retention; Compliance; Orthodontic; Periodontal Health
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive electronic reminder (Experimental): Participants in the intervention group will receive tailored electronic reminders. The frequency and content of the reminders will be informed by the qualitative findings of an ongoing trial, but are likely to include an intra-oral photograph taken pre-treatment and following removal of the active appliances, instructions on the necessary duration of retention, advice on maintenance of retainers, departmental details, advice on appropriate management for appliance breakages, and delineation of the implication of suboptimal retainer wear. Also, information related to the debond visit and maintenance of optimal oral hygiene levels will be incorporated in the mobile application.
  Interventions: Other: Electronic reminder
- Control group (No Intervention): Participants in the control group will not receive additional reminders.

INTERVENTIONS:
Other: Electronic reminder — The frequency and content of the reminders will be informed by the qualitative findings of an ongoing trial, but are likely to include an intra-oral photograph taken pre-treatment and following removal of the active appliances, instructions on the necessary duration of retention, advice on maintenance of retainers, departmental details, advice on appropriate management for appliance breakages, and delineation of the implication of suboptimal retainer wear. Also, information related to the debond visit and maintenance of optimal oral hygiene levels will be incorporated in the mobile application.
  Arms: Receive electronic reminder

SUMMARY:
Participants will be recruited for inclusion at a routine adjustment appointment prior to planned removal of the appliances. Following removal of the appliances, consenting participants will be randomly allocated to one of two groups by computer-generated random allocation. Allocation will be concealed from the treating clinician using of an opaque sealed envelope system. Standard stone model records will be available for all participants following removal of the appliances (T0).

Participants in both groups will have follow-up scheduled for 3 (T1), 6 (T2) and 12 (T3) months following removal of the braces. All participants will be instructed to wear standard clear, plastic (Essix-type) retainers on a full-time basis for 6 months, followed by night-time wear for a further 6 months. A micro-electronic timer will be integrated within the upper Essix-type retainer. All participants will be given standard advice at each recall visit.

Participants in the intervention group will receive tailored electronic reminders in the form of a mobile application. The frequency and content of the reminders will be informed by qualitative interviews involving participants from an allied trial, and from posts related to orthodontic retainers shared on social media. Instructions on the necessary duration of retention, maintenance of retainers, departmental details, allied to advice on appropriate management for appliance breakages, and delineation of the implication of suboptimal retainer wear will be included. Also, information related the debond visit and maintenance of optimal oral hygiene levels will be incorporated in the mobile application. Participants in the control group will not receive additional reminders. Treating clinicians will be kept blind to the study group.

All patients failing an appointment will be sent another. Those wishing to withdraw from the trial may do so at any point without affecting continuing care with records taken at the point of withdrawal from the study with data analysis on an intention to treat basis.

Thereafter, patient experiences with electronic reminders will be evaluated on a subset of participants using one-to-one interviews.

DETAILED DESCRIPTION:
Details related to the intervention:

Participants in the intervention group will receive access to the 'My Retainers' mobile application via a unique identification code. The researcher will demonstrate the use of the mobile application with a brief description of its features. Participants in the control group will not have access to the mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 21 years
* Planned for removable retention with Essix-type vacuum-formed retainers
* In the permanent dentition

Exclusion Criteria:

* Inability to access or peruse electronic mail
* Cleft lip and palate and other craniofacial anomalies

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padhraig Fleming, Study Chair — Queen Mary University of London
Locations (1):
- The Royal London Hospital Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be freely available to reviewers in future and may be made available on a public database

REFERENCES:
- [Derived] Zhang X, Al-Moghrabi D, Pandis N, Shah S, Fleming PS. The effectiveness of a bespoke mobile application in improving adherence with removable orthodontic retention over 12 months: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2022 Mar;161(3):327-337. doi: 10.1016/j.ajodo.2021.09.010. Epub 2021 Nov 17. PMID 34801348
- [Derived] Al-Moghrabi D, Pandis N, McLaughlin K, Johal A, Donos N, Fleming PS. Evaluation of the effectiveness of a tailored mobile application in increasing the duration of wear of thermoplastic retainers: a randomized controlled trial. Eur J Orthod. 2020 Nov 3;42(5):571-579. doi: 10.1093/ejo/cjz088. PMID 31799628

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Events that occurred after enrollment, but prior to assignment of participants to the treatment groups: failure to collect retainers (n= 2); mobile application did not work (n= 1); and sensor deactivated in error (n= 1).
Period: Overall Study
Arm/Group | Receive Electronic Reminder | Control Group
Started | 42 | 42
Completed | 29 | 25
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receive Electronic Reminder | Control Group | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.24 (2) | 17.2 (1.89) | 17.23 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 21 | 21 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Wear of Removable Retainer Per Day (Hours) in the Intervention and the Control Groups
Description: Objective levels of retainer wear will be recorded from an integrated micro-electronic sensor in the retainer
Time Frame: 3 months - 6 months - 12 months
Measure: Median (Standard Error); unit: hours/day
Arm/Group | Receive Electronic Reminder | Control Group
Number analyzed (Participants) | 29 | 25
hours/day | 3.09 (8.1) | 1.44 (9.22)

2. Secondary Outcome: Self-reported Hours of Retainer Wear Per Day
Description: Subjective levels of retainer wear as reported by participants using retainer wear chart
Time Frame: 3 months - 6 months - 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Study Model Based Outcomes
Description: Stability of teeth following orthodontic treatment measured from study models (in millimetres)
Time Frame: 3 months - 6 months - 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Patients' Experience With Electronic Reminders in a Related Qualitative Element (Positive and Negative Experiences, in Addition to Feedback From Participants in Relation to Tailored Electronic Reminders Based on One-to-one Interviews)
Description: Questionnaire
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Assessment of Oral Hygiene Levels and Periodontal Outcomes Including: Plaque Scores, Bleeding on Probing, and Clinical Attachment Level
Description: Clinical assessment
Time Frame: Baseline - 3 months - 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Knowledge With Orthodontic Retainers
Description: Questionnaire
Time Frame: 3 months
Reporting Status: Not Posted

7. Secondary Outcome: Experience With Orthodontic Retainers
Description: Questionnaire
Time Frame: 3 months - 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Anxiety Levels on the Day of Debond
Description: Questionnaire
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of study of 24 months
Description: No harms were observed
Arm/Group | Receive Electronic Reminder | Control Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03224481/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT03224481/ICF_001.pdf